CLINICAL TRIAL: NCT07194837
Title: The Efficiency of 810 nm Diode Laser on Periapical Healing After Root Canal Retreatment Using Cone Beam Computed Tomography: A Randomized Controlled Clinical Trial
Brief Title: The Efficiency of 810 nm Diode Laser on Periapical Healing After Root Canal Retreatment
Acronym: Retreatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Sabah Morad Sobhy, Endodontic department, al azhar university. principal investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-PD-25-27
Record Dates: First submitted 2025-09-19; First posted 2025-09-26 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: This Study Will be Performed to Evaluate the Efficiency of 810 nm Diode Laser Disinfection on Periapical Healing in Root Canal Retreatment Cases
Keywords: disinfection; retreatment; 810 diode laser
MeSH Terms: interventions — Lasers, Semiconductor; Calcium Hydroxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Diode laser group) (Experimental): Laser activated disinfection will be performed using 810 nm diode laser (Elexxion clarosdental laser, Singen Deutschland, Germany) in a continuous wave mode with a power of 1.5 Watts in 4 cycles of 5 seconds with 20 seconds intervals in between each. Prior to irradiation, all the individuals in the room will wear protective laser safety eye glasses. A 200 μm fiber optic tip (Lite medics, Italy) will be inserted 1 mm from the working length, activated and moved in slow helical motion from the apex to the cervical third with alternating between clockwise and counterclockwise direction at speed of about 2 mm/s(23). 5 ml saline solution will be used for each application and finally before tooth restoration temporarily with light cure glass ionomer resin cement.
  After 1 week, the temporary filling will be removed following local anaesthesia and isolation, the root canal will be irrigated with 5 ml saline. Then, the root canal system will be obturated using ADSEAL resin-based
  Interventions: Device: diode laser
- Group II (Calcium hydroxide group) (Experimental): Calcium hydroxide paste (MetaBiomed, Chungcheongbuk-do, Korea) will be placed inside the root canal and left for 1 week. The access cavity will be temporarily sealed with light cure glass ionomer resin cement. After 1 week, the temporary filling will be removed following local anaesthesia and isolation, the root canal will be irrigated with 20 ml saline and gently filed using H file corresponding to the master apical file size. Root canal obturation and final coronal restoration will be completed as in group I.
  Interventions: Other: Calcium Hydroxide (Ca(OH)2)

INTERVENTIONS:
Device: diode laser — 810 nm diode laser (Elexxion clarosdental laser, Singen Deutschland, Germany) in a continuous wave mode with a power of 1.5 Watts in 4 cycles of 5 seconds with 20 seconds intervals in between each.
  Arms: Group I (Diode laser group)
Other: Calcium Hydroxide (Ca(OH)2) — Calcium hydroxide paste (MetaBiomed, Chungcheongbuk-do, Korea) will be placed inside the root canal and left for 1 week.
  Arms: Group II (Calcium hydroxide group)

SUMMARY:
The main cause of endodontic disorders is microbial infection. From the infected root canal, microorganisms can penetrate into the deeper layers of root dentine and propagate a periapical tissue through the apical foramen and lateral canals. Eliminating microorgnims is the primary objective of endodontics in order to create an environment as free of bacteria as possible. This will favor the environment for healing without the need of periapical surgery in some resistant cases.

Disinfection in root canal retreatment (RCR) is much more difficult because persistent microorganisms have settled in the root canal. The resistant periapical lesions result from resistant bacteria to antimicrobial agents. They can survive for years around the filled root canals. Sodium hypochlorite (NaOCl) is the most widely used irrigant in root canal therapy due to its strong antibacterial effect and its ability to dissolve organic substances. Effective canal cleaning is difficult to achieve without the use of NaOCl at a sufficiently high concentration. However, NaOCl has several drawbacks, including its cytotoxicity which can lead to tissue damage and patient symptoms. Additionally, its strong oxidizing nature negatively affects the mechanical properties of dentin such as microhardness and elastic modulus. NaOCl should be used with caution in endodontic procedures to prevent hypochlorite accidents.

Calcium hydroxide (Ca (OH)2) is the most widely utilized intracanal medication. It has the potential to dissolve tissue, acts as a physical barrier and generates hydroxyl ions, creating an extremely alkaline environment. It has been shown to be quite effective in the treatment of teeth with persistent periapical lesions. To provide optimal endodontic treatment, the root canal system should be thoroughly cleaned of soft-tissue debris, smear layer, and bacteria. However, it is impossible to completely disinfect and clean debris that build up. That is why, adjunctive aids, such as the use of passive ultrasonic and sonic activation of the irrigant and lasers with varying wave lengths, have been introduced during conventional endodontic therapy in cleaning maneuvers.

[ Laser therapy for root canal disinfection has gained popularity since laser-assisted root canal treatment aims to remove the smear layer, penetrate deep into dentin and eliminate bacteria up to 1000 μm . Laser types have been shown to reduce bacterial load when used as an adjunct to conventional root canal treatment such as Nd:YAG , Er:YAG and diode laser . Diode laser exhibits a powerful antibacterial effect by altering the bacterial cell wall and damaging the cell membrane. Its photothermal action targets accessible bacteria, while its photodisruptive properties affect those in less accessible areas. This mechanism may not cause immediate bacterial death but instead induces sublethal damage that inhibits bacterial growth. By compromising the integrity of the cell wall and causing the accumulation of denatured proteins, bacterial growth is halted, eventually leading to cell lysis. These effects are achieved with minimal does of heat . Researches have demonstrated differing degrees of effectiveness in achieving root canal disinfection with the use of diode lasers.

Diode laser is highly well-suited for root canal therapy due to its infrared wavelength and the use of a thin, flexible optic fiber tip (200 µm), which enables deep penetration into the root canal system. This design allows for efficient delivery and distribution of laser energy, improving disinfection and reducing microbial load. Furthermore, the compact size and affordability of diode lasers make them practical for use in general dental clinics and increasing their adoption in routine endodontic procedures. A study demonstrated that 980nm diode laser achieved bactericidal effect ranging from 77 to 97% in root canals infected with E. faecalis using energy outputs of 1.7, 2.3 and 2.8 W. Antimicrobial effect was related to the amount of energy and dentin thickness. Furthermore, several studies have confirmed that diode laser can serve as an adjunct to conventional root canal therapy in cases with necrotic pulp and periapical radiolucency because of the bactericidal effect, the ability to penetrate through the dentinal thickness, and the ability to vaporize soft tissues .

Radiographic examination provides essential information on post-treatment periapical healing, where the absence of periapical radiolucency remains a primary marker of successful therapy. Intraoral digital periapical radiograph remains the most widely used imaging modality in endodontics due to their accessibility and reliability. These radiographs provide valuable insights into dentoalveolar structures, allowing clinicians to assess root morphology, canal anatomy, and quality of the treatment. However, the primary limitation lies in its two-dime

DETAILED DESCRIPTION:
Cone beam computed tomography (CBCT) has become a cornerstone in endodontic imaging, providing high-resolution, three-dimensional visualization of complex anatomical structures. CBCT enhances diagnostic precision and treatment planning beyond what is achievable with two-dimensional radiograph. It has been shown to be more accurate than digital periapical radiographs in the long-term assessment of root canal treat¬ment success. Moreover, CBCT demonstrates high accuracy in determining the volume of periapical pathosis making it a valuable tool in periapical healing evaluation. Therefore, this study aims to evaluate the effect of 810 nm diode laser on periapical healing after root canal retreatment in failed endodontic cases with chronic periapical lesion using CBCT. The null hypothesis is that there is no difference in periapical healing between the tested groups following root canal retreatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients have single rooted teeth with root canal form type I.
* Have previous endodontic therapy with failure.
* Have periapical radiolucency (PAI score of 3 or 4).
* Patients who provide written informed consent.

Exclusion Criteria:

* Patients who had received antibiotic therapy within the past month.
* Pregnancy and lactation.
* Systemic disease.
* Physical or mental disability.
* Non restorable teeth.
* Any signs of resorption, immature roots, fracture, perforation.
* Bone metabolism disease and/or patients using drugs that affect bone metabolism (such as steroids and bisphosphonates)

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
periapical healing at 1 year follow-up | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sabah M Sobhy, PHD, Principal Investigator — Al-Azhar University; Eman M. Hassan, Study Director — Faculty of Dental Medicine for Girls, Al-Azhar University, Cairo, Egyp
Locations (1):
- from the outpatient clinic of Endodontic Department, Faculty of Dental Medicine for Girls, Al-Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dogan MU, Aricioglu B, Kose TE, Cikman AS, Oksuzer MC. Association between the irrigation-agitation techniques and Periapical Healing of large periapical lesions: a Randomized Controlled Trial. Clin Oral Investig. 2024 Jun 15;28(7):376. doi: 10.1007/s00784-024-05758-4. PMID 38878107
- [Background] Morsy DA, Negm M, Diab A, Ahmed G. Postoperative pain and antibacterial effect of 980 nm diode laser versus conventional endodontic treatment in necrotic teeth with chronic periapical lesions: A randomized control trial. F1000Res. 2018 Nov 15;7:1795. doi: 10.12688/f1000research.16794.1. eCollection 2018. PMID 31372210